CLINICAL TRIAL: NCT03843749
Title: Pyrotinib in Combination With Trastuzumab in Treatment-refractory, HER2-positive Metastatic Colorectal Cancar.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Zhan Wang, Pyrotinib in Combination With Trastuzumab in Treatment-refractory, HER2-positive Metastatic Colorectal Cancar., Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTHMC
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Cancer
Keywords: HER2; Pyrotinib; Trastuzumab; Metastatic Colorectal Cancar
MeSH Terms: conditions — Colorectal Neoplasms | interventions — pyrotinib; Trastuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HER2-positive Metastatic Colorectal Cancar (Experimental)
  Interventions: Drug: Pyrotinib

INTERVENTIONS:
Drug: Pyrotinib — Pyrotinib in Combination With Trastuzumab
  Other Names: Trastuzumab

SUMMARY:
This clinical trial aims to evaluate the efficacy, safety of Pyrotinib in combination with trastuzumab in Treatment-refractory, HER2-positive Metastatic Colorectal Cancar.

ELIGIBILITY:
Inclusion Criteria:

Patients should be histologically diagnosed with metastatic colorectal cancer or postoperative recurrence; Patients with ALK mutation(including mutation, fusion, rearrangements ); Patients have measurable lesions; Patients are not available for targeted therapy or patients refuse to receive targeted therapy afer second-line treatment; Over 3 weeks after radiotherapy and the radiotherapy focus was not be measured; Age should be 18-25 years; Performance status should be 0-2; Life expectancy should be more than 12 weeks;

Exclusion Criteria:

Patients underwented major surgery or severe trauma within 4 weeks; Patients allergiced to experimental drugs; Patient ready to give birth or who is pregnant; Patients with brain metastases; Patients with chemotherapy contraindication; Patients could not tolerate chemotherapy; Patients have secondary primary tumor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | up to 36 months
  Evaluation of tumor burden based on RECIST criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes